CLINICAL TRIAL: NCT02065999
Title: Surveillance for Antiviral Resistant Variants in Chronic Hepatitis C Patients
Acronym: SEARCH-C
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: VHCRP1107
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C, chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored serum and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-centre prospective longitudinal cohort study with the aim of collecting and storing clinical data, patient blood, DNA and PBMCs to examine outcomes related to drug resistance, drug monitoring and host genetics in the era of directly acting antiviral drugs for hepatitis C therapy.

DETAILED DESCRIPTION:
1. To analyse for resistance-associated HCV variants in DAA-naïve HCV patients using population and ultra-deep pyrosequencing (UDPS). Resistance associated variants will be analysed by qualitative and quantitative methods both pre-treatment and on-treatment.
2. To determine whether in the absence of drug pressure there is variation in the prevalence of naturally occurring resistance associated variants.
3. To correlate the presence and frequency of baseline resistance-associated variants with the response to therapy with DAA-based triple therapy regimens for HCV.
4. To identify predictors of emergent DAA resistance and treatment failure during therapy with DAA-based combination strategies, including virological, clinical and immunological factors.
5. To characterize the natural history of HCV resistance associated variants that are selected during antiviral therapy after the withdrawal of treatment.
6. To establish a cohort of DAA-treatment failure patients suitable for re-treatment studies.
7. To establish a tissue repository of serum and PBMCs from well-characterized patients treated with DAA-based triple therapy to allow future examination of the role of other variables that may potentially impact on the outcomes of DAA based therapy and development of RAVs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection
* Commencing or expected to commence DAA-based HCV treatment within the next year
* IFN treatment-naïve or IFN treatment-experienced
* Provision of written, informed consent

Exclusion Criteria:

* In the opinion of the investigator that the patient is not able to provide informed consent
* Inability or unwillingness to comply with study collection requirements

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated 100 participants will be recruited from 2 study sites: St Vincent's Hospital, Sydney; St Vincent's Hospital, Melbourne.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of HCV resistance associated variants (RAVs) and the incidence of RAVs arising during therapy. | Baseline
  Descriptive statistics will be used to describe RAVs using standard international nomenclature and presented in table form. Baseline clinical and demographic data on subjects will be presented, as will rates of treatment failure and reasons for failure.

SECONDARY OUTCOMES:
Factors associated with treatment failure due to virological breakthrough / relapse. | Baseline
  Multivariable logistic regression modelling with backwards elimination will be used to identify factors associated with this.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Dr Matthews, MBChB, MRCP (UK), FRACP, PhD, Principal Investigator — The University of New South Wales
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - St Vincent's Hospital, Melbourne, Victoria